CLINICAL TRIAL: NCT07019259
Title: Light Therapy for Chemotherapy Induced Peripheral Neuropathy in Childhood Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Rally Foundation for Childhood Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000038498
Record Dates: First submitted 2025-05-23; First posted 2025-06-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Childhood Cancer; Chemotherapy-induced Peripheral Neuropathy
Keywords: Survivors of childhood cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Light Therapy (Experimental): Week 1 will include a baseline evaluation in clinic. In weeks 1-6, participants will complete 18 total light therapy sessions (3 sessions/week, 15/minutes session). The first session will be observed in clinic at the time of the baseline evaluation, and the remaining 17 sessions will be completed at home. In Week 7 survivors will follow-up in clinic for a repeat evaluation with the physical therapist (or study team member). .
  Interventions: Device: Anodyne Therapy System

INTERVENTIONS:
Device: Anodyne Therapy System — Survivors will be provided the Anodyne Therapy System Model 120 to use as part of a 6-week at-home light therapy intervention. Participants will be instructed on where apply the device based on location of their symptoms, and will be instructed to use the device for 15 minutes per day, 3 days per week. Proper use of the device will be demonstrated in clinic by a trained physical therapist or study team member.

SUMMARY:
The purpose of this study is to determine feasibility and acceptability of a six-week at-home light therapy protocol in childhood cancer survivors, to identify facilitators and barriers to implementing this intervention, and to measure signs and symptoms of Chemotherapy Induced Peripheral Neuropathy (CIPN) at baseline and following completion of the at-home light therapy protocol.

DETAILED DESCRIPTION:
This prospective single-arm pilot study will assess the feasibility of a 6-week at-home light therapy intervention for CIPN. Survivors of childhood cancer (<21 years at diagnosis), ages five years or older at the time of survivorship clinic visit, with a history of exposure to vinca alkaloid, platinum, or other chemotherapeutic agent that can cause CIPN, will be included if they have CIPN (defined as a score of four or higher on the pediatric modified Total Neuropathy Score for survivors <18 years old at evaluation, or the modified Total Neuropathy Score for survivors 18 years or older at evaluation). The primary outcome of the study will be feasibility of the at-home protocol, measured as proportion of survivors who complete at least 12 at-home light therapy sessions, with ≥70% of survivors completing 12 or more sessions indicating feasibility. Secondary outcomes include 1) Proportion of survivors satisfied with intervention, measured as a mean score of 3 or higher on a 4-point Likert-scale survey 2) Facilitators and barriers to implementation of light-therapy, assessed by semi-structured qualitative interviews with 5-10 survivors who adhered and did not adhere to the protocol, and 3) change in neuropathy symptoms (measured by change in modified Total Neuropathy Score or pediatric-modified Total Neuropathy Score, and gait speed) from baseline to 1 week post intervention.

ELIGIBILITY:
Inclusion Criteria:

* History of childhood cancer (<21 years of age at diagnosis)
* Current age five years or older (due to availability of validated measures for CIPN in this age group)
* History of exposure to vinca alkaloid, platinum, or other chemotherapeutic agent that can cause CIPN
* CIPN as assessed by a trained physical therapist defined as a score of four or higher on the ped-mTNS (for survivors <18 years old at evaluation), or the mTNS (for survivors 18 years or older at evaluation)

Exclusion Criteria:

* Currently Pregnant or lactating (by patient report, at initiation or at any point of the study)
* Inability to sit still for at least 15 minutes
* Diagnosis of neuropathy prior to cancer treatment
* Active cancer diagnosis or cancerous skin lesion
* Central nervous system tumor (due to lack of validated measures for CIPN in this population)
* Cancer lesion or open wound in the area to be treated, or any condition that can potentially be made worse by the correct or incorrect use of the device.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of light therapy protocol | 7 weeks
  Measured as proportion of participants adhering to protocol (completing 12 of 18 sessions), with ≥70% of participants adhering to the protocol indicating feasibility

SECONDARY OUTCOMES:
Acceptability of light therapy for CIPN | 7 weeks
  Proportion of participants reporting satisfaction with the intervention, measured by a participant survey assessing satisfaction on a 4-point Likert scale (1-very dissatisfied, 2-somewhat dissatisfied, 3-somewhat satisfied, 4-very satisfied), total score range 1-4 with a mean score of 3 or higher indicating satisfaction.
Barriers and facilitators | 7 weeks
  List of perceived barriers and facilitators to the intervention derived from qualitative interviews.
Change in gait efficiency | baseline and 7 weeks
  Measured by change in 6-minute walk distance from baseline to completion of the intervention. It measures the distance an individual can walk over a total of six minutes on a hard, flat surface.
Changes in neuropathy symptoms | baseline and 7 weeks
  Measured by the pediatric modified Total Neuropathy Score (ped-mTNS for survivors <18 years old) and the modified Total Neuropathy Score (mTNS, for survivors 18 years or older) from baseline to completion of the intervention. For ped-mTNS the total score ranges from 0 to 32, with higher scores indicating more severe neuropathy. For ped-mTNS the total score ranges from 0 to 24, with higher scores indicating more severe neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Rozalyn Rodwin, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Health Smilow York Street Hospital, New Haven, Connecticut
  - Yale New Haven Health Park Avenue Medical Center, Trumbull, Connecticut

IPD SHARING:
Plan to Share IPD: No